CLINICAL TRIAL: NCT04504786
Title: Effects of the Vitality Acupunch Exercise Program on the ADL and Functional Fitness of Sarcopenia Older Adults
Brief Title: Vitality Acupunch Exercise Program for Sarcopenia Older Adults
Acronym: VA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Kuei-Min Chen, Ph.D., RN., Professor, Kaohsiung Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KMUHIRB-F(II)-20190045(1)
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Activities of Daily Living; Functional Fitness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitality acupunch (VA) (Experimental): The VA program took 40 minutes to complete and included three phases: 1) activating qi and blood (5 movements, 10 minutes): warm-up exercises that allowed the body to accumulate heat and promote flexibility of the joints to loosen up the body, 2) punching meridians (14 movements, 20 minutes): both hands were used to exert a vibrating effect according to the rhythms that stimulate the 14 meridians in the entire body to improve aerobic endurance, and 3) relaxing body and mind (5 movements, 10 minutes): muscle relaxing exercises to rest the body and cease the qi. Participants in the experimental group received the VA program led by the instructors, who were trained and certified by the PI, 3 times per week and 40 minutes per session for 6 months.
  Interventions: Other: Vitality acupunch (VA) exercise program
- Control (Active Comparator): Participants in the control group continued with their daily activities as usual.
  Interventions: Other: Control

INTERVENTIONS:
Other: Vitality acupunch (VA) exercise program — The VA had three phases and took 40 minutes to complete.
  Arms: Vitality acupunch (VA)
Other: Control — Participants maintained their daily activities.
  Arms: Control

SUMMARY:
This project was aimed to test the effects of a six-month VA program on the activities of daily living (ADL) and functional fitness of institutional older adults with sarcopenia.

DETAILED DESCRIPTION:
A cluster-randomized controlled trial was conducted to test the effects of a six-month VA program on ADL and functional fitness (lung capacity, body flexibility, range of the joint's motion, and muscle endurance) of institutional older adults with sarcopenia. Using convenience sampling, 12 long-term care facilities with 114 older adults were recruited, and then cluster-randomized by the facility to a VA experimental or a control group. The experimental group received the VA program led by certified instructors 3 times per week and 40 minutes per session for six months; the control group continued with their regular daily activities. One pre-test and two post-tests, three months apart, were conducted.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 65 years old
* have been living in the facility for at least three months
* intact cognitive function with the Short Portable Mental Status Questionnaire (SPMSQ) score ≥ 8
* hand-grip strength < 28 kg for men and < 18 kg for women
* calf circumference < 34 cm for men and < 33 cm for women

Exclusion Criteria:

* have spinal cord injury
* have severe cardiovascular or pulmonary diseases
* have musculoskeletal diseases

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 114 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2021-03-06 (Actual); Study Completion 2021-03-06 (Actual)

PRIMARY OUTCOMES:
Lung capacity | 6 months
  measured by the TruZoneTM Peak Flow Meter
Upper body flexibility | 6 months
  measured by the Back Scratch Test
Lower body flexibility | 6 months
  measured by the Chair Sit-and-Reach Test
Range of joint motion | 6 months
  measured by the goniometry
Arm muscle endurance | 6 months
  measured by the Arm Curl Test
Leg muscle endurance | 6 months
  measured by the Chair-to-Stand Test

SECONDARY OUTCOMES:
Activities of daily living (ADL) | 6 months
  measured by the Barthel Index. The score of "0-20" means totally dependent; "21-60" means heavily dependent; "61-90" means moderately dependent; "91-99" means mildly dependent; "100" indicates total independence in the ADL of a person.

CONTACTS AND LOCATIONS:
Overall Officials: Kuei-Min Chen, PhD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tung HT, Chen KM, Huang KC, Hsu HF, Chou CP, Kuo CF. Effects of Vitality Acupunch exercise on functional fitness and activities of daily living among probable sarcopenic older adults in residential facilities. J Nurs Scholarsh. 2022 Mar;54(2):176-183. doi: 10.1111/jnu.12723. Epub 2021 Nov 8. PMID 34751506